CLINICAL TRIAL: NCT00612976
Title: Symbicort in Chronic Obstruktive Pulmonary Disease
Acronym: SYMBIOSE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Kai Richter, AstraZeneca Germany
Other Study IDs: 1312006001; budesonide /formoterol; German PMS trial no.8
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: treatment of COPD; documentation of relevant data; related to the budesonide/formoterole therapy in patients with COPD.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with COPD treated with budesonide/formoterol

SUMMARY:
Under daily routine conditions and without any intervention by the sponsor regarding the selection of subjects, diagnostic procedures, therapeutic decisions (medicinal and non- medicinal therapy, dose, duration, etc.), routine assessments, the participating physicians (i.e.general practitioners and internists) are asked to document relevant data related to the budesonide/formoterole therapy in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD treated with budesonide/formoterol

Exclusion Criteria:

* limitiations; possible risks; warnings; contraindications mentioned in the SPC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general practitioners and internists
Sampling Method: Probability Sample
Enrollment: 18014 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
efficacy and tolerability of budesonide /formoterole in subjects with COPD who are treated by general practitioners and internists. | change of a quality of life score compared to baseline by using CRQ, stratified by present therapy and severity of COPD; incidence of the occurrence of unknown, unexpected and/or rarely occurring adverse events AE under outpatient medical care conditions

SECONDARY OUTCOMES:
to get further insight into the details of the use , dosage scheme and duration of treatment with budesonide /formoterol in this population

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Chair — Medical Department AstraZeneca Germany